CLINICAL TRIAL: NCT04558229
Title: Randomized Control Trial Evaluating Impact of Standardized Counseling on Early Discontinuation for Irregular Bleeding in Users of the Contraceptive Implant
Brief Title: RCT Evaluating Standardized Counseling on Early Discontinuation for Irregular Bleeding in Nexplanon Users
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Planned Parenthood of the St. Louis Region and Southwest Missouri (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MSD201959528
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Birth Control; Contraception; Contraceptive Usage; Family Planning
Keywords: Contraceptive implant; Birth control; Nexplanon
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: 1:1 fashion with block sizes of 8 using a computer-generated random allocation
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study team members will be blinded to the randomization, with the exception of the research member who will be delivering the counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Clinician Counseling (No Intervention)
- Additional Standardized Counseling (Experimental)
  Interventions: Other: Additional Standardized Counseling

INTERVENTIONS:
Other: Additional Standardized Counseling — Research staff will follow a script designed to give unbiased, medically accurate information regarding bleeding changes that may occur with use of a contraceptive ENG implant.
  Arms: Additional Standardized Counseling

SUMMARY:
Clinician counseling for implant users should involve an explanation of the likelihood of irregular bleeding and the possibility of continued or frequent bleeding throughout three years of use. If that counseling does not provide specifics of the actual distribution of bleeding patterns described in published literature, there remains the real possibility of biased or directed counseling, leading to an inaccurate and exaggerated expectation of potential bleeding changes. This study aims to evaluate if a standardized script accompanied by a visual aid regarding expected bleeding profiles, with intention to remove any possibility of negative or positive framing, could change users' expectations and satisfaction with their method, leading to lower discontinuation rates.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at the health center to receive an etonogestrel-releasing subdermal implant (Nexplanon) for primarily contraceptive benefits
* Ability to consent in English

Exclusion Criteria:

* Have used an etonogestrel-releasing subdermal implant (Nexplanon) within the 12 weeks prior to enrollment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-gendered females; Assigned female at birth and not using hormone therapy
Enrollment: 348 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Nexplanon Discontinuation Rates | 6 months
  Based subjects' self-reported ability to cope with various changes in bleeding patterns, and other demographic information, we will analyze whether an association exists between those who discontinue their method use early due to troublesome bleeding and the counseling they received on the day of method insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen P McNicholas, DO, MSCI, Principal Investigator — Planned Parenthood of the St. Louis Region and Southwest Missouri
Locations (1):
- Planned Parenthood of the St. Louis Region and Southwest Missouri, St Louis, Missouri, United States